CLINICAL TRIAL: NCT02222675
Title: Comparison of Sonographically Assisted With Conventionally Breast Surgery - Prospective, Randomised, Multicenter, Parallel Group Study With Two Study Arms
Brief Title: Conserving Breast Surgery - Comparison of Conventional With Sonography
Acronym: MAC-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Women's Hospital Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MAC-001_1.1
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Breast Surgery

ARMS (2):
- Sonographically assisted breast surgery (Experimental): Sonographically assisted breast surgery
  Interventions: Procedure: Sonography assisted breast surgery
- Conventional breast surgery (Active Comparator): Conventional breast surgery
  Interventions: Procedure: Conventional breast surgery

INTERVENTIONS:
Procedure: Sonography assisted breast surgery
  Arms: Sonographically assisted breast surgery
Procedure: Conventional breast surgery
  Arms: Conventional breast surgery

SUMMARY:
Aim of the study is to test whether surgical removal of a tumor under sonographic control as compared to conventional method reduces the rate of resections and local relapse

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years
* Female
* Presurgical validated breast cancer

Exclusion Criteria:

* Sonographically not defined report
* Lobular breast cancer
* Extensive ductal carcinoma in situ

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-04; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Rate of second tumor resections | Five years

CONTACTS AND LOCATIONS:
Locations (1):
- University Women's Hospital, Tübingen, Germany

REFERENCES:
- [Derived] Hoffmann J, Marx M, Hengstmann A, Seeger H, Oberlechner E, Helms G, Rohm C, Ott C, Wallwiener D, Stabler A, Wiesinger B, Hartkopf AD, Brucker SY, Hahn M. Ultrasound-Assisted Tumor Surgery in Breast Cancer - A Prospective, Randomized, Single-Center Study (MAC 001). Ultraschall Med. 2019 Jun;40(3):326-332. doi: 10.1055/a-0637-1725. Epub 2018 Jul 5. PMID 29975969